CLINICAL TRIAL: NCT01761565
Title: Single- and Multiple-Dose Pharmacokinetics of Sublingual Sufentanil NanoTab® PCA System (Zalviso™) in Healthy Subjects
Brief Title: Single and Multiple Dose Pharmacokinetics of Sufentanil NanoTab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Talphera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IAP101
Record Dates: First submitted 2013-01-03; First posted 2013-01-07 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Plasma Concentrations
MeSH Terms: interventions — Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single dose of SUF NT 15 mcg then 40 doses of SUF NT 15 mcg (Experimental): Period 1: Single dose of SUF NT 15 mcg
  Period 2: 40 consecutive doses of SUF NT 15 mcg taken every 20 minutes
  Interventions: Drug: Single dose of SUF NT 15 mcg; Drug: 40 consecutive doses of SUF NT 15 mcg taken every 20 minutes

INTERVENTIONS:
Drug: Single dose of SUF NT 15 mcg
Drug: 40 consecutive doses of SUF NT 15 mcg taken every 20 minutes
  Other Names: Zalviso™

SUMMARY:
Determine the plasma concentration profile after single and multiple dosing of Sufentanil NanoTabs

ELIGIBILITY:
Inclusion Criteria:

* Non smoking
* Ages 18 to 45 year, inclusive
* BMI between 18 and 30

Exclusion Criteria:

* Subjects taking any prescription or OTC medications or vitamins or supplements
* Pregnant females
* Subjects with pulmonary disease or sleep apnea

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra K. Willsie, D.O., Principal Investigator — PRA
Locations (1):
- PRA, Lenexa, Kansas, United States

REFERENCES:
- [Background] Willsie SK, Evashenk MA, Hamel LG, Hwang SS, Chiang YK, Palmer PP. Pharmacokinetic properties of single- and repeated-dose sufentanil sublingual tablets in healthy volunteers. Clin Ther. 2015 Jan 1;37(1):145-55. doi: 10.1016/j.clinthera.2014.11.001. Epub 2014 Dec 24. PMID 25544247

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Dose of SUF NT 15 mcg Then 40 Doses of SUF NT 15mcg: Arm 1/Period 1: Single dose of SUF NT 15 mcg
  Subjects received oral naltrexone 50 mg approximately 14 and 2 hours before and 10 hours after the SUF NT dosing
  Arm 2/Period 2: 40 consecutive doses of SUF NT 15 mcg
  Subjects received oral naltrexone 50 mg approximately 2 hours before and 10, 22, and 34 hours after the first dose of SUF NT in Period 2.
Period: Single Dose of SUF NT 15 mcg
Arm/Group | Single Dose of SUF NT 15 mcg Then 40 Doses of SUF NT 15mcg
Started | 40
Completed | 40
Not Completed | 0
Period: 40 Consecutive Doses of SUF 15 mcg
Arm/Group | Single Dose of SUF NT 15 mcg Then 40 Doses of SUF NT 15mcg
Started | 39 (Subject was withdrawn from the study prior to the second arm/period due to non-compliance)
Completed | 38
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: One patient was withdrawn after Period 1 due to non-compliance
Groups:
- One Dose of SUF NT 15 mcg Then 40 Doses of SUF NT 15 mcg: Arm 1/Period 1: Single dose of SUF NT 15 mcg
  Single dose of SUF NT 15 mcg
  Arm 2/Period 2: 40 consecutive doses of SUF NT 15 mcg
  40 consecutive doses of SUF NT 15 mcg
Arm/Group | One Dose of SUF NT 15 mcg Then 40 Doses of SUF NT 15 mcg
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: For Treatment A, serial blood samples were taken at 0 (predose), 5, 10, 15, 20, 30, 40, 50, 60, 70, 80, 90, 120, 180, 240, 360, 480, 600, 720, 800, and 840 minutes, and 24 hours after the Sufentanil NanoTab dose on Day 1.
  For Treatment B, serial blood samples were collected at 0, 20, 120, 240, 360, 480, 600, 720, 760, 780, 785, 790, 795, 800, 810, 820, 830, 840, 850, 860, 870, 900, 960, 1020, 1140, 1260, 1380, 1500, 1580, and 1620 minutes, and 37 hours after the first Sufentanil NanoTab dose on Day 3
Time Frame: 24 hours in Treatment A, 37 hours in Treatment B
Population: 2 of the 40 subjects had incomplete PK data and were excluded from PK analysis (1 due to early withdrawal and 1 due to AE)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Single Dose of SUF NT 15 mcg | 40 Consecutive Doses of SUF NT 15 mcg
Number analyzed (Participants) | 38 | 38
pg/mL | 34.96 (12.23) | 249.55 (72.13)

2. Primary Outcome: Time to Steady State
Description: Steady state, for the cohort, was assessed using Helmert's method (ratio of the geometric mean concentration of each time point to the geometric mean concentrations pooled over all remaining time points, and achieved at the first not-statistically significant time point (i.e., p >0.05)
Time Frame: 24 hours
Population: as for outcome 1
Measure: Number; unit: hours
Arm/Group | 40 Consecutive Doses of SUF NT 15 mcg
Number analyzed (Participants) | 38
hours | 4

3. Primary Outcome: CST½
Description: the time for plasma concentrations to decrease from Cmax to 50% of Cmax after discontinuation of drug administration
Time Frame: 24
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Groups:
- Single Dose of SUF NT 15 mcg: Arm 1/Period 1: Single dose of SUF NT 15 mcg
Arm/Group | Single Dose of SUF NT 15 mcg | 40 Consecutive Doses of SUF NT 15 mcg
Number analyzed (Participants) | 38 | 38
hours | 2.17 [0.17 to 5.00] | 2.66 [1.33 to 3.95]

ADVERSE EVENTS:
Time Frame: AEs were collected from administration of the first dose of study drug through completion of the post-treatment procedures.
Arm/Group | Single Dose of SUF NT 15 mcg | 40 Consecutive Doses of SUF NT 15 mcg
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 5/40 | 18/39
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Dose of SUF NT 15 mcg (N=40) | 40 Consecutive Doses of SUF NT 15 mcg (N=39)
Photophobia (Eye disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 6
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Feeling abnormal (General disorders) | 0 | 1
Feeling jittery (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 6
Somnolence (Nervous system disorders) | 0 | 4
Dizziness (Nervous system disorders) | 0 | 3
Syncope vasovagal (Nervous system disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hot flush (Vascular disorders) | 0 | 3
Flushing (Vascular disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 — All adverse events listed in the above table are included regardless of relationship to study drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must be able to review any publications prior to publication